CLINICAL TRIAL: NCT04173533
Title: A Double-Blind, Phase III, Randomised Study to Compare the Efficacy and Safety of Oral Azacitidine (CC-486) Versus Placebo in Subjects With Acute Myeloid Leukaemia or Myelodysplastic Syndromes as Maintenance After Allogeneic Haematopoietic Stem Cell Transplantation
Brief Title: Randomised Study of Oral Azacitidine vs Placebo Maintenance in AML or MDS Patients After Allo-SCT
Acronym: AMADEUS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RG_18-048
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Acute Myeloid Leukemia; Myelodysplasia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — Azacitidine; cc-486

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Oral azacitidine (CC-486) matched placebo once daily for first 14 days of each 28 day cycle
  Interventions: Drug: Matched placebo
- Experimental Group (Experimental): Oral azacitidine (CC-486) 200 mg once daily for first 14 days of each 28 day cycle
  Interventions: Drug: Oral azacitidine

INTERVENTIONS:
Drug: Oral azacitidine — Oral azacitidine (CC-486) 200 mg tablet
  Other Names: CC-486
  Arms: Experimental Group
Drug: Matched placebo — Oral azacitidine (CC-486) matched placebo tablet
  Other Names: Oral azacitidine matched placebo
  Arms: Control Group

SUMMARY:
This study will evaluate a new maintenance therapy with the aim of improving the outcome of patients with acute myeloid leukaemia (AML) and myelodysplasia (MDS) after stem cell transplantation.

DETAILED DESCRIPTION:
This is a prospective, two arm, double-blind, phase III clinical trial in adult patients with acute myeloid leukaemia (AML) and myelodysplasia (MDS) who have undergone an allogeneic stem cell transplant (allo-SCT) and are randomised to receive oral azacitidine or placebo upon engraftment for up to 12 months as maintenance therapy. Patients will be stratified by type of transplant (myeloablative/reduced intensity, age (<60/≥ 60 years) and donor type (sibling/unrelated)).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 16 at the time of signing the informed consent form
2. Patients with a diagnosis of any of the below:

   * AML (CR1 or CR2) according to World Health Organization (WHO) classification;
   * Secondary AML (defined as previous history of MDS, antecedent hematological disease or chemotherapy exposure; CR1 or CR2); or
   * Advanced or high risk MDS with an IPSS-R of ≥3.5 (intermediate 3.5 or higher) including intermediate or high risk chronic myelomonocytic leukaemia (CMML) (e.g. CPSS int-2 or high risk) (as per IPSS-R)

   undergoing allo-SCT using myeloablative conditioning (MAC) or reduced-intensity conditioning (RIC) preparative regimens, and with either peripheral blood or bone marrow as the source of hematopoietic stem cells.
3. At the time of allo-SCT

   * No prior allo-SCT; and
   * No more than 1 antigen mismatch at HLA-A, -B, -C, -DRB1 or -DQB1 locus for either related or unrelated donor; and
   * No haplotype or cord blood donor; and
   * Bone marrow blast <5% for AML and <10% for MDS patients
4. Able to commence therapy between 42 to 84 days following allo-SCT
5. Post-transplant bone marrow

   1. AML patients - blast count ≤ 5% confirmed within 28 days prior to starting study therapy
   2. MDS patients - confirmation of CR post-transplant with blast count ≤ 5% in bone marrow
6. Adequate neutrophil and platelet engraftment within 14 days prior to starting study therapy defined as:

   * Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L on two consecutive testing without daily use of myeloid growth factor; and
   * Platelet ≥ 50 x 10^9/L on two consecutive testing without platelet transfusion within 1 week
7. Adequate organ function:

   * Serum aspartate aminotransferase (AST) and alanine transaminase (ALT) < 4 x upper limit of normal (ULN)
   * Serum bilirubin < 2 x ULN. Higher levels are acceptable if these can be attributed to active red blood cell (RBC) precursor destruction within the bone marrow (i.e., ineffective erythropoiesis) or Gilbert's syndrome
   * Serum creatinine < 2 x ULN
8. Adequate coagulation (Prothrombin time (PT) ≤ 15 seconds and partial thromboplastin time (PTT) ≤ 40 seconds)
9. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
10. Patients with adequately controlled GVHD (defined as GVHD grade <II with concurrent use of corticosteroids equivalent of prednisone at a dose ≤ 0.5 mg/kg) can be included
11. Females of childbearing potential (FCBP) may participate, providing they meet the following conditions:

    1. Agree to use at least two effective contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomised partner) or practice true abstinence throughout the study, and for 6 months following the last dose of study therapy and
    2. Have a negative serum pregnancy test (sensitivity of at least 25 mIU/mL) at screening; and
    3. Have a negative serum or urine (investigator's discretion) pregnancy test (sensitivity of at least 25 mIU/mL) within 72 hours prior to starting study therapy. This applies even if the subject practices complete abstinence from heterosexual contact.
12. Male patients with a female partner of childbearing potential must agree to the use of at least two physician-approved contraceptive methods throughout the course of the study and should avoid fathering a child during the course of the study and for 3 months following the last dose study therapy
13. Understand and voluntarily sign an informed consent from prior to any study related assessments or procedures being conducted
14. Able to adhere to the study visit schedule (i.e., clinic visits at the study sites are mandatory, unless noted otherwise for study visits) and other protocol requirements

Exclusion Criteria:

1. Use of any of the following after transplantation and prior to starting study therapy:

   * Any chemotherapy used for adjuvant therapy
   * Unlicensed investigational agents/therapies used within 28 days prior to starting study therapy
   * Azacitidine, decitabine or other hypomethylating agent (HMA)
   * Lenalidomide, thalidomide and pomalidomide used within 28 days prior to starting study therapy
2. Subjects who have undergone a haploidentical or cord blood transplant
3. Active GVHD grade II or higher (acute GVHD Clinical Staging and Grading)
4. Concurrent use of corticosteroids equivalent of prednisone at a dose > 0.5 mg/kg
5. Known active viral infection with Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV)
6. Active uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment)
7. History of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis), celiac disease (i.e., sprue), prior gastrectomy or upper bowel removal, or any other GI disorder or defect that may interfere with the absorption, distribution, metabolism or excretion of the investigational medicinal products (IMPs) and/or predispose the subject to an increased risk of gastrointestinal toxicity prior to allo-SCT
8. Idiopathic thrombocytopenic purpura (ITP), disseminated intravascular coagulation, haemolytic uremic syndrome, thrombotic thrombocytopenic purpura (TTP)
9. History of prior malignancies, except: lobular breast carcinoma in situ, fully resected basal cell or squamous cell carcinoma of skin or treated cervical carcinoma in situ, Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, node, metastasis (TNM) clinical staging system), previous MDS, CMML, myeloproliferative neoplasms (MPN) resulting in secondary AML. Cancer treated with curative intent ≥ 5 years previously will be allowed. Cancer treated with curative intent < 5 years previously will not be allowed.
10. Significant active cardiac disease within the previous 6 months, including:

    * New York Heart Association (NYHA) class III or IV congestive heart failure
    * Unstable angina or angina requiring surgical or medical intervention; and/or
    * Myocardial infarction
11. Known or suspected hypersensitivity to azacitidine or mannitol
12. Pregnant or lactating females
13. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from participating in the study.
14. Any condition including the presence of laboratory abnormalities, which places the patient at unacceptable risk if he/she were to participate in the study
15. Any condition that confounds the ability to interpret data from the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Relapse free survival (RFS) | 12 months
  To determine RFS at one year from randomisation of oral azacitidine compared with placebo in patients undergoing allo-SCT for AML/MDS

SECONDARY OUTCOMES:
Overall survival (OS) | 12 and 24 months
  OS at one and two years from randomisation of oral azacitidine compared with placebo
Cumulative incidence of relapse (CIR) | 12 and 24 months
  CIR at one and two years after treatment comparing oral azacitidine with placebo
Non-relapse mortality (NRM) | Day 100 and 12 months
  NRM at 100 days and 12 months after treatment comparing oral azacitidine with placebo
Incidence of acute and chronic graft-versus-host disease (GVHD) | 24 months
  Incidence of acute and chronic GVHD comparing oral azacitidine with placebo
Time to early treatment discontinuation | 24 months
  Time to early treatment discontinuation comparing oral azacitidine with placebo
Safety (adverse events) | 24 months
  Number of patients with adverse events on oral azacitidine compared with placebo
Quality of Life (EORTC-QLQ-C30 and EQ-5D) | 24 months
  QoL will be measured to compare oral azacitidine with placebo
GVHD-free and relapse-free survival (GRFS) | 12 and 24 months
  GRFS defined as time from date of randomisation to date of first event or death

CONTACTS AND LOCATIONS:
Overall Officials: Charles Craddock, Principal Investigator — University of Birmingham
Locations (20):
- United Kingdom (20):
  - The Queen Elizabeth Hospital, Birmingham
  - University Hospital Bristol, Bristol
  - Addenbrooke's Hospital, Cambridge
  - University Hospital of Wales, Cardiff
  - Queen Elizabeth University Hospital, Glasgow
  - St. James's University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Clatterbridge Cancer Centre, Liverpool
  - Hammersmith Hospital, London
  - King's College Hospital, London
  - St Bartholomew's Hospital, London
  - The Royal Marsden Hospital, London
  - University College London Hospitals, London
  - Manchester Royal Infirmary, Manchester
  - The Christie Hospital, Manchester
  - Freeman Hospital, Newcastle
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No